CLINICAL TRIAL: NCT05181163
Title: In Vitro Biofilm Formation and Antibiotic Susceptibility Patterns of Bacteria From Surgical Site Infection After Orthopedic Surgery
Brief Title: Biofilm Formation and Antibiotic Sensitivity Patterns
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Ahmed Talaat, Principal investigator, Sohag University
Other Study IDs: Soh-Med-21-11-03
Record Dates: First submitted 2021-12-08; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Orthopedic Surgery
Keywords: biofilm antibiotics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: swab — Swabs from site of infection will be taken

SUMMARY:
Detection of bacteria that form biofilm and its sensitivity to antibiotics in patients with surgical site infection after orthopedic surgery.

DETAILED DESCRIPTION:
The available number of patients presenting in outpatient clinic or at operating theatre with surgical site infection after orthopedic surgery that include insertion of implant (e.g plates , screws ,wires ,…) will be subjected to full history and examined by physician. Swabs from site of infection will be taken and subjected to the following steps to identify the causative bacteria:

* Culturing on blood agar, chocolate agar, MacConkey agar and Mannitol salt agar , gram staining and biochemical tests.
* Enzyme-linked immunosorbent assay (ELISA) to detect biofilm formation.
* Antimicrobial Susceptibility Testing using the Kirby-Bauer disk diffusion method.

ELIGIBILITY:
Inclusion Criteria:

* patients with surgical site infection after orthopedic surgery that include insertion of implant (e.g plates , screws ,wires ,…)

Exclusion Criteria:

* if patient has no orthopedic surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients presenting in outpatient clinic or at operating theatre with surgical site infection after orthopedic surgery that include insertion of implant (e.g plates , screws ,wires ,…)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
detect biofilm formation | one year
  The available number of patients presenting in outpatient clinic or at operating theatre with surgical site infection after orthopedic surgery that include insertion of implant (e.g plates , screws ,wires ,…) will be subjected to full history and examined by physician. Swabs from site of infection will be taken and subjected to Enzyme-linked immunosorbent assay (ELISA) to detect biofilm formation.

CONTACTS AND LOCATIONS:
Overall Officials: principal investigator, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided